CLINICAL TRIAL: NCT01522638
Title: Cross Sectional Study of Autosomal Dominant Opticus Atrophy
Brief Title: Advanced Characterization of Autosomal Dominant Optic Atrophy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Cecilia Rönnbäck, MD, Glostrup University Hospital, Copenhagen
Other Study IDs: ADOA
Record Dates: First submitted 2011-11-30; First posted 2012-01-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Optic Atrophy, Autosomal Dominant
MeSH Terms: conditions — Optic Atrophy, Autosomal Dominant

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADOA: This group includes subjects diagnosed with autosomal dominant optic atrophy
- Healthy subjects

SUMMARY:
The purpose of this study is to determine the anatomy of the retina and the optic nerve in patients with autosomal dominant optic atrophy (ADOA). Based on these findings the aim of the study is to determine why patients with the same type of genetic material, i.e. the same mutation, have such large variations of symptoms, spanning from unaffected subjects to blindness. The project requires examination of both healthy and affected family members.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with autosomal dominant optic atrophy

Exclusion Criteria:

* Age below 8 years old

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with autosomal dominant optic atrophy in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 1 day
vessel caliber | 1 day
OCT | 1 day
Microperimetry | 1 day
Lifestyle questionnaire | 1 day
General checkup | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael Larsen, MD, Prof. DMSc, Principal Investigator — Glostrup University Hospital
Locations (1):
- Copenhagen University, Glostrup Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Ronnback C, Larsen M. Macular sensitivity and fixation patterns in patients with autosomal dominant optic atrophy. Dan Med J. 2014 Sep;61(9):A4888. PMID 25186535